CLINICAL TRIAL: NCT03465683
Title: Transmission of ESBL-producing Enterobacteriaceae and Their Mobile Genetic Elements-identification of Sources by Whole Genome Sequencing
Brief Title: Transmission of ESBL-producing Enterobacteriaceae
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00100; me18Tschudin
Record Dates: First submitted 2018-03-01; First posted 2018-03-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hospital Acquired Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Enterobacteriaceae
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ESBL-producing Enterobacteriaceae — Data and biological sample collection

SUMMARY:
The aim of this research project is to investigate the transmission of ESBL-producing Enterobacteriaceae on both, the level of bacterial strains and mobile genetic elements, and to determine the source of hospital-acquired infections.

DETAILED DESCRIPTION:
Background and aim The most common bacterial pathogens in humans include several species of the family of Enterobacteriaceae. Many of them have now become resistant to antibiotics, i.e.extended-spectrum beta-lactamases (ESBL)-producing Enterobacteriaceae (PE). For a long time it was thought that transmission in hospitals was the main factor driving their rapid spread. More recently, though, ESBL-PE have also been found on food and in waste water. These sources are also likely to play an important role in entertaining transmission.

Investigator's aim is to identify transmission chains of ESBL-PE in the Basel urban region, using the latest whole genome sequencing methodologies allowing to determine relatedness of strains with the highest possible resolution, taking into account sources both within and outside hospitals.

Hypothesis The finding of few genetically-related clusters of ESBL-PE with an epidemiological link to hospital contacts would suggest relevant transmission in our healthcare setting. In contrast, the finding of many genetically-distinct clusters of ESBL-PE without epidemiological links to the hospital, would question the importance of hospital-wide transmission in sustaining the ESBL epidemic. This distinction is critical for deriving effective prevention and control recommendations.

Design, setting and patients Whole genome sequencing will be performed on representative ESBL-strains collected from January 2003 to December 2019 at the University Hospital Basel. The epidemiological relationships between patients with genetically related strains of ESBL-PE will be assessed.

From June 2017 to December 2019, whole genome sequencing will in addition be performed on ESBL-strains identified from representative samples from the wastewater system of both the hospital and the city of Basel as well as representative foodstuff samples collected from both the hospital and the city of Basel. The epidemiological relationships between patients, as well as environmental samples with genetically related strains of ESBL-PE and cases with genetically related plasmids carrying the respective ESBL genes will be assessed.

Methods, planned analysis and sample size To identify transmission events we will employ whole genome sequencing with Illumina technology, which is established and International Standards Organization (ISO)-accredited at the Clinical Microbiology Department at the University Hospital. The proportion of infection/colonization with genetically related isolates of ESBL-producing Enterobacteriaceae of the overall infection/colonization rate will be determined. All phylogenies will be inferred using BEAST v2.046 employing our previously developed tool for quantifying transmission rates. Overall, 2000 isolates from patient's samples and 1000 isolates from food and wastewater samples will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* aged above 1 year
* proven ESBL-PE carriage from any specimens obtained by routine clinical practice out and inpatients from University Hospital Basle from January 1st until December 31st 2019

Exclusion Criteria:

* not meeting inclusion criteria

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: out and inpatients from University Hospital Basle
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection/colonization proportion | through study completion, an average of 45months
  The proportion of infection/colonization with genetically related isolates of ESBL-producing Enterobacteriaceae (primary outcome) of the overall infection/colonization rate will be determined and stratified for both, in and outpatient setting for species and time periods

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tschudin-Sutter, PD MD, Principal Investigator — Division of Infectious Disease and Hopital Epidemiology, University Hospital Basle
Locations (1):
- University Hospital Switzerland, Division of Infecteous Disease and Hospital Epidemiology, Basel, Switzerland

REFERENCES:
- [Derived] Aguilar-Bultet L, Bagutti C, Egli A, Alt M, Maurer Pekerman L, Schindler R, Furger R, Eichenberger L, Roloff T, Steffen I, Huebner P, Stadler T, Tschudin-Sutter S. Identification of a Cluster of Extended-spectrum Beta-Lactamase-Producing Klebsiella pneumoniae Sequence Type 101 Isolated From Food and Humans. Clin Infect Dis. 2021 Jul 15;73(2):332-335. doi: 10.1093/cid/ciaa1164. PMID 32776135